CLINICAL TRIAL: NCT01898975
Title: Evaluation of Stroke Volume Variation Derived From NICOM as a Predictor of Fluid Responsiveness in Neurosurgical Patients: A Gray Zone Approach
Brief Title: A Gray Zone Approach to Stroke Volume Variation Derived From NICOM
Status: Withdrawn | Type: Observational
Why Stopped: The investigators decided not to proceed this study because of some internal matters.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-03-053-001
Record Dates: First submitted 2013-06-28; First posted 2013-07-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Neurological Diseases or Conditions; Fluid Responsiveness; Non Invasive Cardiac Output Monitoring; Gray Zone
Keywords: Neurosurgical patients; Fluid loading; Fluid responsiveness; NICOM; Stroke volume variation; Pulse pressure variation; Total peripheral resistance; Gray zone approach

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 500ml fluid loading: All enrolled patients
  Interventions: Other: 500ml fluid loading

INTERVENTIONS:
Other: 500ml fluid loading — Fluid loading to evaluate fluid responsiveness
  Other Names: 500ml loading of crystalloid(Plasma Solution-A Injection CJ) over 15min; at the end of operation, when the main procedure finished and there is no strong; stimulation with stable hemodynamics

SUMMARY:
Optimal fluid management has been considered as crucial part to determine postoperative outcome and organ function. Recently developed, non invasive cardiac output measurement(NICOM, Cheetah Medical, Portland, OR)has enabled continuous cardiac output(CO) monitoring just by attaching electrode on chest wall. Moreover, CO and SSV derived from NICOM have been demonstrated as predictors of fluid responsiveness. Therefore, the aim of this study is to evaluate stroke volume variation derived from NICOM as a predictor of fluid responsiveness in neurosurgical patients. In addition, we plan to reveal inconclusive patients using gray zone approach.

DETAILED DESCRIPTION:
Optimal fluid management has been considered as crucial part to determine postoperative outcome and organ function. Many reports have focussed on evaluation of fluid responsiveness using various parameters such as pulse pressure variation (PPV) or stroke volume variation (SSV) derived from invasive or semi-invasive monitoring. Recently developed, non invasive cardiac output measurement(NICOM, Cheetah Medical, Portland, OR)has enabled continuous cardiac output(CO) monitoring just by attaching electrode on thorax. Moreover, CO and SSV derived from NICOM have been demonstrated as predictors of fluid responsiveness. Therefore, the aim of this study is to evaluate stroke volume variation derived from NICOM as a predictor of fluid responsiveness in neurosurgical patients. In addition, we plan to reveal inconclusive patients using gray zone approach.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or ASA II patients aged 20-80 undergoing neurosurgery in supine position

Exclusion Criteria:

* Pre-existing arrythmic disorders
* Congestive heart failure required medical treatment
* Preoperative Creatinine 1.3mg/dl
* observing self respiration during the study interventions
* Bleeding tendency
* Severe brain edema

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing neurosurgery under general anesthesia in supine position
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Stroke volume variation | 5min following the end of rapid fluid infusion
  5min following the end of rapid fluid infusion: 5 min after the end of fluid loading

SECONDARY OUTCOMES:
Correlation with pulse pressure variation | 5 min following the end of rapid fluid infusion
  5min following the end of rapid fluid infusion: 5 min after the end of fluid loading

OTHER OUTCOMES:
TPR(total peripheral resistance), TPRI(total peripheral resistance index) | 5min following the end of rapid fluid infusion
  5min following the end of rapid fluid infusion: 5 min after the end of fluid loading

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Hwan Lee, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung medical center, Seoul, South Korea